CLINICAL TRIAL: NCT05034159
Title: A Pilot Trial of CBT-I for Sleep, Pain, and Inflammation in Crohn's Disease
Brief Title: CBT-I for Sleep, Pain, and Inflammation in Crohn's Disease
Acronym: SPIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Crohn's and Colitis Foundation (Other)
Responsible Party: Principal Investigator, Jessica.K.Salwen-Deremer, Principal Investigator, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: STUDY02001191
Record Dates: First submitted 2021-09-01; First posted 2021-09-05 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Crohn Disease; Insomnia; Sleep Disturbance; Pain; Inflammation
MeSH Terms: conditions — Crohn Disease; Sleep Initiation and Maintenance Disorders; Parasomnias; Pain; Inflammation | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Following a baseline assessment, participants are initially randomized to either CBT-I or waitlist. Those in the waitlist condition will repeat their baseline assessment after 8 weeks, then will start CBT-I.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Behavioral Therapy for Insomnia (Experimental): CBT-I has a specific protocol with behavioral targets that differ significantly from standard CBT. This approach focuses on implementing sleep restriction and stimulus control interventions which are fully deployed during the first session. Five CBT-I sessions will be delivered over the course of 8 weeks. Key recommendations include: 1) reduce time in bed; 2) get up at the same time every day; 3) do not go to bed unless sleepy; 4) do not stay in bed awake for more than 15 minutes; and 5) avoid napping. Participants are also taught relaxation strategies and cognitive therapy addresses arousal and catastrophizing.
  Interventions: Behavioral: Cognitive Behavioral Therapy for Insomnia
- Waitlist (No Intervention): No intervention for 8 weeks.

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy for Insomnia — Same as is described previously.
  Arms: Cognitive Behavioral Therapy for Insomnia

SUMMARY:
People with Crohn's disease often suffer from sleep problems. Long term, sleep problems may lead to more flares of Crohn's disease or other complications. In general, people with Crohn's disease also report that sleep problems can worsen symptoms of Crohn's disease the next day. In people with other medical problems, research has also shown that having sleep problems can make other things worse, such as pain and inflammation. In this study, the researchers want to understand the treatment of sleep problems in people with Crohn's disease, and what else might improve if sleep gets better. This study will use Cognitive Behavioral Therapy for Insomnia (CBT-I) to treat insomnia symptoms. CBT-I is the recommended treatment for insomnia and has been shown to improve sleep problems, pain, and inflammation in other groups of people. If this study is successful, it will contribute to understanding how to treat insomnia in people with Crohn's disease and how sleep impacts pain and inflammation. Long term, this information will be helpful in understanding how best to take care of people with Crohn's disease.

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate Crohn's disease (as assessed by PRO-3 score)
* Insomnia severity index score of 8 or greater
* Sleep onset latency and/or wake after sleep onset of at least 30 minutes
* Access to device and internet/cell phone service sufficient for telehealth

Exclusion Criteria:

* PHQ-9 score of 20 or greater
* GAD-7 score of 20 or greater
* Unstable major psychiatric condition
* Current alcohol or substance abuse
* Current narcotic use for pain control
* Current systemic corticosteroid use
* Current pregnancy or nursing
* Ileostomy or colostomy
* Diagnosis of seizure disorder
* Diagnosis of sleep apnea or positive STOP-Bang screen
* Diagnosis of restless leg syndrome or positive Cambridge-Hopkins RLSq screen
* Night shift, rotating shift work, or frequent travel outside of primary time zone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2021-10-22 (Actual); Primary Completion 2023-04-19 (Actual); Study Completion 2023-04-19 (Actual)

PRIMARY OUTCOMES:
Change in insomnia symptoms as measured by the Insomnia Severity Index | From baseline assessment to 1-month post intervention
  The Insomnia Severity Index (ISI) is a self-report questionnaire designed to measure severity of insomnia. The ISI is made up of 7 items on insomnia symptoms and related impairments and total scores range from 0-28. Higher scores are indicative of greater insomnia symptoms.
Change in diary-based sleep onset latency | From baseline assessment to 1-month post intervention
  A weekly average of self-reported time it takes to fall asleep each night, derived from a self-reported sleep diary
Change in diary-based wake after sleep onset | From baseline assessment to 1-month post intervention
  A weekly average of self-reported time spent awake in the middle of each night, derived from a self-reported sleep diary

SECONDARY OUTCOMES:
Change in sleep efficiency based on diary | From baseline assessment to 1-month post intervention
  Change in sleep efficiency (total sleep time / time in bed), derived from a self-reported sleep diary
Change in sleep efficiency based on actigraphy | From baseline assessment to 1-month post intervention
  Change in sleep efficiency (total sleep time / time in bed) as measured by actigraphy (actigraph)
Change in diary sleep efficiency based on ambulatory EEG monitoring | From baseline assessment to 1-month post intervention
  Change in sleep efficiency (total sleep time / time in bed) as measured by ambulatory EEG sleep architecture monitoring (sleep profiler)
Change in sleep onset latency as measured by actigraphy | From baseline assessment to 1-month post intervention
  Change in sleep onset latency as measured by actigraphy (actigraph)
Change in wake after sleep onset as measured by actigraphy | From baseline assessment to 1-month post intervention
  Change in wake after sleep onset as measured by actigraphy (actigraph)
Change in sleep onset latency as measured by ambulatory EEG monitoring | From baseline assessment to 1-month post intervention
  Change in sleep onset latency as measured by ambulatory EEG sleep architecture monitoring (sleep profiler)
Change in wake after sleep onset as measured by ambulatory EEG monitoring | From baseline assessment to 1-month post intervention
  Change in wake after sleep onset as measured by ambulatory EEG sleep architecture monitoring (sleep profiler)
Change in self-reported pain as measured by the Brief Pain Inventory | From baseline assessment to 1-month post intervention
  The Brief Pain Inventory will be used to assess pain location, severity, and interference. Pain severity is rated from 0-10 and pain interference is rated from 0-10; higher scores indicate more severe pain and more pain interference.
Change in behaviorally assessed pain tolerance via the Cold Pressor Test | From baseline assessment to 1-month post intervention
  The Cold Pressor Test involves submerging one's non-dominant hand in ice water and rating discomfort at regular, pre-determined intervals. Pain tolerance will be measured based on the total amount of time a participant can keep their hand submerged, with a maximum of 2 minutes.
Change in self-reported Crohn's disease symptoms as measured by the Patient Reported Outcomes-3 | From baseline assessment to 1-month post intervention
  The Patient Reported Outcomes-3 is a self-report questionnaire that assesses frequency of diarrhea, severity of abdominal pain, and overall well-being. Higher scores indicate more severe Crohn's disease symptoms.
Change in time spent in slow wave sleep | From baseline assessment to 1-month post intervention
  We will measure percentage of time spent in slow wave sleep during a night's sleep using the Sleep Profiler, an ambulatory EEG sleep monitor
Change in C-reactive protein | From baseline assessment to 1-month post intervention
  We will measure blood levels of C-reactive protein
Change in fecal calprotectin | From baseline assessment to 1-month post intervention
  We will measure levels of fecal calprotectin via a stool sample.

CONTACTS AND LOCATIONS:
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No